CLINICAL TRIAL: NCT04230226
Title: A Randomized, Double-blind, Placebo Controlled, Single-center Study to Determine the Effects of Pre-workout and Recovery Formulations on Soreness, Performance, Tolerance and Safety Outcomes in Healthy Adults Undergoing Training Program
Brief Title: Acute Study on Muscle Soreness, Damage, and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 20-PHX-0001 Acute
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Soreness, Muscle; Performance Enhancing Product Use; Damage Muscle
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-workout and Post-workout Product (Active Comparator): Pre-workout plus: a blend of caffeine, choline bitartrate, carbohydrate, HMB, vitamin D3 mixed with water and consumed within 30 minutes prior to exercise
  Protein recovery plus: a blend of whey protein, caseinate, carbohydrate, vitamin C, alpha-tocopherol, vitamin D3, glucosamine mixed with water and consumed 15 minutes post exercise
  Interventions: Dietary Supplement: Pre-workout plus and protein recovery plus
- Study Placebo (Placebo Comparator): non-caloric powder mixed with water consumed within 30 minutes prior to exercise and within 15 minutes post exercise
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pre-workout plus and protein recovery plus — Study products consumed prior and after exercise
  Arms: Pre-workout and Post-workout Product
Other: Placebo — Placebo product consumed prior and after exercise
  Arms: Study Placebo

SUMMARY:
The acute study will evaluate pre- and post-exercise ingestion of a multi-ingredient supplement in a randomized, double-blind, placebo-controlled, crossover design. Participants will complete one enrollment visit, in which they will sign a consent form and complete a health history questionnaire. Participants will complete two interventions, with three visits each (6 visits total), in which a treatment beverage (pre/post supplement, or non-caloric placebo) will be consumed within 30 minutes prior to exercise and within 15 minutes post-exercise, in random order. Total time from enrollment to completion will be at least 14 days. Testing visits will be separated by a minimum of 7 days of rest to allow for recovery and washout, based on a half-life of ≤8 hours for all ingredients present in the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Participant is an adult between the ages of 25-50 years
* Participant has a recorded BMI of 20-35 kg/m2
* Participant exercises less than 3 hours per week for at least 8 weeks preceding the study
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing to and able to comply with the protocol
* Participant is apparently healthy and no reported metabolic disorders, heart disease, arrhythmias, thyroid disease, renal, hepatic, autoimmune or neurological diseases, as determined by a health history questionnaire
* Participant agrees to maintain current diet and exercise routine during the study
* Participant agrees to refrain from taking any anti-inflammatory supplement 48 hours prior to exercise (acute) or medications to prevent any further nutritional or drug related protection against exercise induced muscle damage
* Participant has a resting (seated for 5 minutes) blood pressure of systolic pressure between 140-90 mmHg and a diastolic pressure between 90-50 mmHg

Exclusion Criteria:

* Participant is currently enrolled in a separate clinical trial or weight loss program involving diet, exercise, physical activity, or the potential ingestion of an active drug or dietary supplement
* Participant is using, or has consistently used one of the following dietary supplements within 12 weeks prior to enrollment: Beta-alanine, Creatine, HMB, Carnosine, Vitamin D
* Participant has consistently consumed whey protein/plant protein and/or 1,000 mg of fish oil within the previous 4 weeks prior to enrollment
* Participant has gained or lost ≥ 8 lbs in the previous month
* Participant has a known allergy or sensitivity to the placebo or active ingredients
* Participant has used tobacco more than three days per week (on average) in the previous 6 months, or refuses to abstain from all tobacco use for the duration of the study
* Participant is pregnant or planning to become pregnant
* Participant has any musculoskeletal condition prohibiting them from participation

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Performance | baseline, 24 hours, 48 hours
  Change from baseline on performance by measuring countermovement vertical jump height using a jump mat and associated velocity using a linear transducer.

SECONDARY OUTCOMES:
Muscle soreness | baseline, 24 hours, 48 hours
  Change from baseline on muscle soreness using visual analog scale (a horizontal 100 mm line where zero will represent no soreness and one-hundred will represent maximum amount of soreness. Participants will be asked to place a single vertical that represents their current soreness. The scale will be measured with a calibrated ruler with the higher numbers representing more soreness.)
Creatine Kinase | baseline, 24 hours, 48 hours
  Change from baseline on muscle damage by measuring creatine kinase
Isoprostanes | baseline, 24 hours, 48 hours
  Change from baseline on muscle damage by measuring isoprostanes

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No